CLINICAL TRIAL: NCT02245685
Title: Longitudinal Followup of Patients Under Substitution Therapy From the Moment They Enter a Specialized Care Center for Addicts to the Period They Are Monitored by a General Practitioner Outside the Specialized Care Center
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: French Health Products Safety Agency (Other Government)
Responsible Party: Sponsor
Other Study IDs: BRD/07/07-M
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Addiction
Keywords: Substitution Therapy; Specialized Care Center for Addicts
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is part of the french priorities of the 2007-2011 addiction plan. Priority #2 of the plan underlines the need to improve practices and access to opioid substitution treatment. Priority 3 stresses the importance of articulation and coordination between specialized structures and community medicine to optimize the quality of care and to ensure continuity in the followup of these patients. This study focuses on the followup of patients under substitution therapy from the moment they enter a specialized care center for addicts to the period they are monitored by a general practitioner outside the specialized care center. The assessment described in this study should allow to harmonize and keep a continuity in patient monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients entering a specialized medical care center for addicts

Exclusion Criteria:

* Patients refusing to sign the consent for participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients under substitution therapy monitored in a specialized care center for addicts
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2008-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Evolution of the severity score to heroin addiction (TMSP score) | From the time patients start to be followed in the specialized care center to the time they leave the specialized care center (up to 5 years)

SECONDARY OUTCOMES:
Evolution of the score of quality of life scale | From the time patients start to be followed in the specialized care center to the time they leave the specialized care center (up to 5 years)
Evolution of the severity score to heroin addiction (TMSP score) | From the time patients leave the specialized care center to the time they are followed by a general practitioner (up to 5 years)
Evolution of the score of quality of life scale | From the time patients leave the specialized care center to the time they are followed by a general practitioner (up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Pascale JOLLIET, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- CSST "La Rose des Vents", Saint-Nazaire, France

REFERENCES:
- [Derived] Guillou-Landreat M, Levassor P, Guerlais M, Sebille V, Victorri-Vigneau C. Prospective Study on Factors Associated with Referral of Patients with Opioid Maintenance Therapy from Specialized Addictive Disorders Centers to Primary Care. Int J Environ Res Public Health. 2021 May 27;18(11):5749. doi: 10.3390/ijerph18115749. PMID 34071908